CLINICAL TRIAL: NCT05370469
Title: Real-Time Monitoring and Modeling of Symptoms and Adverse Events in Lung Cancer Patients Receiving Oral Targeted Therapies for Tumors With Actionable Mutations
Brief Title: Real-Time Monitoring of Symptoms in Lung Cancer Patients Receiving Oral Targeted Therapies
Acronym: Lung001
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Ryan Gentzler, MD, Principal Investigator, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSR210257
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer; EGFR Gene Mutation; EGFR; ALK Gene Mutation; RET Gene Mutation; MET Gene Mutation; KRAS Mutation-Related Tumors; BRAF; ROS1 Gene Mutation
Keywords: EGFR gene mutation; EGFR; ALK; Fitbit; Tyrosine kinase inhibitor; TKI; Fitbit Sense; Sensus; RX Cap; Smart pill cap; Smart cap; Smartphone; Smartwatch; Fitness watch; Remote monitoring; survey; RET mutation; MET mutation; KRAS mutation; BRAF mutation; ROS1 mutation
MeSH Terms: conditions — Lung Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Subjects who, at enrollment, have been on a TKI for less than 4 weeks will be monitored with the Sensus smartphone application, Fitbit Sense, RX Cap, and paper surveys. Visits will be at: Screening, Baseline, 1 Week, 2 Weeks, 4 Weeks, 8 Weeks, 16 weeks, and 24 weeks.
  Interventions: Other: Sensus Smartwatch Application; Device: RX Cap; Device: Fitbit Sense; Other: Surveys
- Cohort B (Experimental): Subjects who, at enrollment, have been on a TKI for 4 weeks or more will be monitored with the Sensus smartphone application, Fitbit Sense, RX Cap, and paper surveys. Visits will be at: Screening, Baseline, Week 1, and then every 8 weeks for 24 weeks.
  Interventions: Other: Sensus Smartwatch Application; Device: RX Cap; Device: Fitbit Sense; Other: Surveys

INTERVENTIONS:
Other: Sensus Smartwatch Application — Sensus is capable of administering ecological momentary assessments (EMAs) on a schedule, randomly, or using sensor-triggers. In this way, Sensus will capture both active (patient-initiated) and passive data streams from native smartphone sensors. Passive streams may include, but are not limited to, GPS, accelerometer, gyroscope, and pedometer data. Participants will be able to log data such as their activity, symptoms and medication adherence via user-initiated surveys within the Sensus app. Sensus will also prompt users to record their medication adherence, symptoms, or activity. This will be done either at fixed intervals (e.g., three times daily) or whenever the onboard sensors detect potential changes in a user's physiological state (e.g., shaking / moving around).
Device: RX Cap — The RXCap medication event monitoring device will be used to collect data on participant adherence to their TKI medication. A small computer chip is included in the top of a pill bottle. When the cap is taken off of the pill bottle by turning it or unscrewing it, the cap records the time and date that it was removed.
Device: Fitbit Sense — The Fitbit Sense smartwatch will be used to collect data including steps, calories burned, total distance travelled, sleep (e.g. time spent sleeping and quality of sleep), flights of stairs climbed, active minutes, exercise (e.g. minutes spent exercising at various intensities), and average heart rate.
Other: Surveys — Electronic and paper surveys will be administered throughout the study.

SUMMARY:
In this study, patients who are taking oral tyrosine kinase inhibitor (TKI) therapy for lung cancer will be asked to participate in a remote monitoring system for up to 24 weeks. The system will include:

* a smartphone application (app) developed at the University of Virginia called Sensus. Sensus will be downloaded to the participant's smartphone. The app will collect active data (such as through surveys) and passive data (such as accelerometer data).
* a fitness watch called a Fitbit will be given to the participant to be used during the study. The Fitbit will collect information such as steps and average heart rate.
* a smart pill cap called RX Cap will be given to the participant to be used during the study. The pill cap will collect information about how often a pill bottle is opened.

The study will also involve paper surveys that are taken by the participant during clinic visits. Symptoms related to TKI therapy will be recorded by an investigator in the clinic.

The study results will be used to guide development of a real-time symptom monitoring system, with the ultimate goal of improving TKI symptom response and quality of life.

DETAILED DESCRIPTION:
This is a prospective pilot study for adult patients with lung cancer who have tumors harboring an actionable mutation and who are undergoing treatment with oral tyrosine kinase inhibitors (TKIs). The choice and dose of TKI will be at the discretion of the treating medical oncologist. The study will assess symptoms and adverse events using a remote monitoring system that uses brief self-report surveys and passive input from smart devices as well as clinical assessment of adverse events and quality of life during routine office visits. An application loaded onto a smart phone (Sensus) and a fitness tracking device (Fitbit Sense) will capture information about symptoms and adverse events. This information will be captured through surveys and from passive input from the smart devices. Surveys will also be used to capture the subjects' experience with the devices. The results of this pilot study will be used to guide future development of a mobile health system application for remote real-time symptom monitoring to implement earlier interventions to reduce severity of symptoms, improve quality of life, and avoid drug discontinuations and dose reductions in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, ≥18 years of age
* Diagnosis of non-small cell lung cancer (NSCLC) with an actionable mutation
* Currently prescribed oral tyrosine kinase inhibitors (TKIs). Participants may or may not have started taking the TKI prior to enrollment on this study. Participants who are initiating TKI treatment or are within 4 weeks of initiation of TKI treatment will be eligible for Cohort A. Participants who have been receiving TKIs for 4 or more weeks will be eligible for Cohort B.
* Owns a smartphone or tablet
* Ability and willingness to download and use a smart device application for the purposes of this study. Ability and willingness to use a Fitbit watch for the purposes of this study.
* Must have the ability to access WiFi or a device with mobile network (3G, 4G, 5G, etc.) connectivity during the course of the study
* Must be English speaking

Exclusion Criteria:

* Any physical or cognitive impairment that would prevent the subject from using the study devices or participate in the study procedures.
* Any ongoing clinically significant grade ≥2 adverse events attributed to a previously prescribed TKI that is a different TKI from the one prescribed at enrollment for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using the remote system to capture symptoms associated with TKI administration. | 24 Weeks
  Number of participants wearing the device and responding to remote electronic surveys at least 50% of the time.

SECONDARY OUTCOMES:
Estimate frequency and severity of adverse events | 24 Weeks
  Adverse event frequency and severity recorded by the app and from in-person clinical assessments using the CTCAE v5.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Gentzler, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No